CLINICAL TRIAL: NCT05265754
Title: The Effect of Sujok Therapy on Pain, Fatigue, Insomnia, Nausea and Vomiting Experienced by Patients With Gastrointestinal System Cancer
Brief Title: The Effect of Sujok Therapy on Cancer Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Demet GUNES, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Demettez
Record Dates: First submitted 2022-02-04; First posted 2022-03-04 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Pain; Insomnia; Fatigue; Nausea and Vomiting; gastrointestinal system cancer.; sujok therapy
MeSH Terms: conditions — Neoplasms; Pain; Sleep Initiation and Maintenance Disorders; Fatigue; Nausea; Vomiting; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: 6 sessions in 2 weeks in total of sujok therapy will be applied to the interventional group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the hand area, firstly, the points will be determined by means of the diagnostic stick and massage will be applied with buckwheat seeds. This massage will be 3 sessions a week, and a total of 6 sessions in 2 weeks.
  Interventions: Behavioral: sujok therapy
- control group (No Intervention): A questionnaire will be applied to the patients by the researcher. Questionnaires will be made as pre-test and post-test.

INTERVENTIONS:
Behavioral: sujok therapy — sujok therapy
  Arms: Experimental group

SUMMARY:
The aim of this study is to determine the effect of Sujok therapy on Pain, Fatigue, Insomnia, Nausea and Vomiting experienced by patients with gastrointestinal system cancer.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of Sujok treatment on Pain, Fatigue, Insomnia, Nausea and Vomiting experienced by patients with gastrointestinal system cancer. Intervention and control groups will be determined by randomization. The scales to be used in the measurement will be applied to the individuals included in the study. Then, sujok therapy will be applied to the intervention group. After 6 sessions in weeks in total, measurement tools will be applied and evaluated again.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Fatigue Severity Measurement - Visual Analogue Scale (VAS) fatigue score of 3 and above,
* Pain Severity Measurement - Visual Analogue Scale (VAS) pain score of 3 and above,
* Measurement of Nausea and Vomiting Severity - Patients with a Visual Analogue Scale (VAS) nausea and vomiting score of 3 and above will be included.

Exclusion Criteria:

* Loss of sensation, amputation, injury, colostomy, etc., which will prevent practice in hands. patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Sujok Therapy's Positive Change in Pain Experienced by Gastrointestinal System Cancer Patients | 2 weeks
  To assess the pain, the MCgill Pain Scale will be applied before starting the sujok application and after the sujok applied for 2 weeks.
Sujok Therapy's positive change in Fatigue Experienced by Patients with Gastrointestinal System Cancer | 2 weeks
  To assess the fatigue, the cancer fatigue scale will be applied before starting the sujok application and after the sujok applied for 2 weeks.
Sujok Therapy's positive cahange in insomnia Experienced by Patients with Gastrointestinal System Cancer | 2 weeks
  In order to evaluate insomnia,the insomnia severity index will be applied before starting the sujok application and after the sujok applied for 2 weeks
Sujok Therapy's positive cahange in nausea and vomiting Experienced by Patients with Gastrointestinal System Cancer | 2 weeks
  To evaluate nausea and vomiting, the Rhodes nausea vomiting scale will be applied before starting the sujok application and after the sujok applied for 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Universty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No